CLINICAL TRIAL: NCT04950946
Title: Natural History of GNAO1-associated Neurodevelopmental Disorder
Brief Title: GNAO1 Natural History Study
Acronym: GNAO1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Bow Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201901128
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: GNAO1
Keywords: Natural History Study; pediatric; neurology; movement disorder; epilepsy; GNAO1
MeSH Terms: conditions — Movement Disorders; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the GNAO1 Natural History Study is to establish the clinical phenotype of GNAO1 associated neurologic disease, its association with genotype, and areas of clinical importance within the disease.

DETAILED DESCRIPTION:
GNAO1 associated neurologic disease is a rare autosomal dominant neurodevelopmental disorder characterized genetically by heterozygous de novo mutations in GNAO1 gene which encodes Gαo, the α subunit of Go, a G protein signal transducer. Phenotypically, it is characterized by developmental delay, epilepsy and/or movement disorder. Medical therapy is symptomatic and often ineffective for many patients. While there are basic and translational studies underway to develop more mechanistic treatments aimed at developing disease modifying treatments, our general knowledge of the natural history of GNAO1 associated neurologicis is extremely limited, making it difficult to select the best measures for identifying changes over time. Without this information,it will be difficult to detect any potential therapeutic efficacy in future trials of novel therapies. To address this critical void in our understanding, we propose to retrospectively and prospectively examine symptom progression(short-and long-term)and developmental outcomes in patients with GNAO1 associated neurologic disease. Retrospective data will be collected on a cohort of 50 patients. Standardized historical clinical information will be received from the physicians and care-givers of these patients, in collaboration with the Bow Foundation Registry. These data will provide an overview of the onset and severity of symptoms over development. In addition, prospective data will be acquired during in-person clinical evaluations of a cohort of 15-20 patients who are not receiving any experimental interventions. In combination, these two approaches will provide critical information about the natural history of GNAO1 associated neurologic disease in children, identify metrics that track change most reliably over time, and collect pilot data for larger future studies.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Bow Foundation GNAO1 registry.
* Evidence of a known pathogenic mutation in GNAO1 or a variant of unknown significance and clinical symptoms likely to be consistent with GNAO1 as determined by study physicians.

Exclusion Criteria:

* Inability to obtain informed consent from parents or adult subjects.
* Inability to obtain medical records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Minors and adults who have a confirmed pathogenic mutation in GNAO1 or a variant of unknown significance and clinical symptoms likely to be consistent with GNAO1 (e.g. global developmental delay, movement disorder, seizures) as determined by study physicians.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Chorea | March 2019; May-Oct 2020
  The Abnormal Involuntary Movement Scale (AIMS) assesses the severity of dyskinesias, as well as the overall severity, incapacitation, and the subject's level of awareness of the movements, and distress associated with them.
Dystonia | March 2019; May-Oct 2020
  The Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) assesses the severity of dystonia in nine body regions. The scale takes into account the severity and frequency of the dystonic movements.
Gross motor development, mobility | March 2019; May-Oct 2020
  The Gross Motor Function Measure (GMFM-88) is a standardized observational instrument designed and validated to measure changes in gross motor function over time in children with cerebral palsy.
Spasticity | March 2019
  The Modified Ashworth Scale (MAS) is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion. The MAS is the current standard for clinical assessment of extremity spasticity.
Fine motor development | March 2019
  The Peabody Developmental Motor Scales 2nd Edition (PDMS-2) is an early childhood motor development program that provides both in-depth assessment and training or remediation of gross and fine motor skills. The assessment is composed of six subtests that measure interrelated motor abilities that develop early in life. We are mainly interested in two subtests: Grasping and Visual-Motor Integration.
Quality of Life and Caregiver Burden | March 2019; May-Oct 2020
  The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) questionnaire attempts to understand and quantitate the quality of life of patients and caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Viehoever, MD, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Ananth AL, Robichaux-Viehoever A, Kim YM, Hanson-Kahn A, Cox R, Enns GM, Strober J, Willing M, Schlaggar BL, Wu YW, Bernstein JA. Clinical Course of Six Children With GNAO1 Mutations Causing a Severe and Distinctive Movement Disorder. Pediatr Neurol. 2016 Jun;59:81-4. doi: 10.1016/j.pediatrneurol.2016.02.018. Epub 2016 Mar 17. PMID 27068059
- [Background] Feng H, Sjogren B, Karaj B, Shaw V, Gezer A, Neubig RR. Movement disorder in GNAO1 encephalopathy associated with gain-of-function mutations. Neurology. 2017 Aug 22;89(8):762-770. doi: 10.1212/WNL.0000000000004262. Epub 2017 Jul 26. PMID 28747448
- [Background] Saitsu H, Fukai R, Ben-Zeev B, Sakai Y, Mimaki M, Okamoto N, Suzuki Y, Monden Y, Saito H, Tziperman B, Torio M, Akamine S, Takahashi N, Osaka H, Yamagata T, Nakamura K, Tsurusaki Y, Nakashima M, Miyake N, Shiina M, Ogata K, Matsumoto N. Phenotypic spectrum of GNAO1 variants: epileptic encephalopathy to involuntary movements with severe developmental delay. Eur J Hum Genet. 2016 Jan;24(1):129-34. doi: 10.1038/ejhg.2015.92. Epub 2015 May 13. PMID 25966631
- [Background] Narayanan UG, Fehlings D, Weir S, Knights S, Kiran S, Campbell K. Initial development and validation of the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD). Dev Med Child Neurol. 2006 Oct;48(10):804-12. doi: 10.1017/S0012162206001745. PMID 16978459
- See also: The Bow Foundation website — https://gnao1.org